CLINICAL TRIAL: NCT02350868
Title: A Phase 1, First-In-Human, Dose-Seeking Study Evaluating the Safety, Pharmacokinetics, and Pharmacodynamics of Orally Administered MPT0E028 in Subjects With Advanced Solid Malignancies Without Standard Treatment
Brief Title: Dose-Seeking Study of MPT0E028 in Subjects With Advanced Solid Malignancies Without Standard Treatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MPT0E028-101
Record Dates: First submitted 2015-01-13; First posted 2015-01-30 (Estimated); Last update posted 2019-04-11 (Actual); Status verified 2018-09

CONDITIONS: Advanced Solid Malignancies
Keywords: without Standard Treatment
MeSH Terms: interventions — 3-(1-benzenesulfonyl-2,3-dihydro-1H-indol-5-yl)-N-hydroxyacrylamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1 (Experimental): Subjects will be treated with oral doses of MPT0E028 in consecutive, 28-day cycles, and will be evaluated regularly for safety. Subjects who tolerate the drug and who do not experience progressive disease may continue to receive MPT0E028 at the discretion of the principal Investigator for up to 6 cycles.
  Interventions: Drug: MPT0E028

INTERVENTIONS:
Drug: MPT0E028 — The starting dose in the Dose Escalation Phase will be 50 mg/day.Dose escalation from the first cohort to the second cohort will be doubled; and from the second cohort to the fourth cohort will proceed at no more than 50% increments.

SUMMARY:
The Dose Escalation Phase will determine the MTD of MPT0E028 and evaluate its safety and tolerability, PK, PD, and preliminary clinical effects; the subsequent Dose Confirmation Phase will be a cohort expansion at or below the MTD (i.e., an RP2D) of MPT0E028.

DETAILED DESCRIPTION:
This is an open-label, non-randomized, dose-escalation study that will evaluate MPT0E028 in subjects with advanced solid malignancies. Subjects will be treated with oral doses of MPT0E028 in consecutive, 28-day cycles, and will be evaluated regularly for safety. Subjects who tolerate the drug and who do not experience progressive disease may continue to receive MPT0E028 at the discretion of the principal Investigator for up to 6 cycles. The Sponsor will keep providing drug for extension cycles to subjects whose disease is controlled at the end of 6th cycle until the end of the study or until the early study termination determined by sponsor. Subjects will return for a follow-up visit 28 days after completion of the end of Study.

ELIGIBILITY:
Inclusion Criteria

1. Males and females ≥ 20 years of age.
2. Pathologically confirmed advanced solid tumor, occurring in progressed disease after treatment with standard therapy, and for which standard therapy proven to provide clinical benefit does not exist.

   NOTE: For primary liver cancer, the standard therapies, such as transcatheter arterial chemoembolization (TACE), radiofrequency ablation (RFA) and percutaneous ethanol intratumor injection (PEI).
3. Eastern Collaborative Oncology Group (ECOG) Performance Status of ≤1 (Appendix 1).
4. Evaluable disease, either measurable on physical examination (PE) or imaging by Response Evaluation Criteria in Solid Tumors (RECIST v1.1, Appendix 4), or by informative tumor marker(s).
5. Laboratory values at screening:

   1. ANC ≥1,500/mm3;
   2. Platelets ≥100,000/mm3;
   3. Total bilirubin ≤1.5 × the upper limit of normal (ULN);
   4. Aspartate aminotransferase (AST [SGOT]) ≤2.5 × the ULN;
   5. Alanine aminotransferase (ALT [SGPT]) ≤2.5 × the ULN;
   6. Serum creatinine ≤1.5 mg/dL or a measured creatinine clearance ≥60 mL/min; and
   7. Negative serum beta- hCG test in women of childbearing potential (defined as women ≤50 years of age or history of amenorrhea for ≤12 months prior to study entry).
6. Subjects with primary liver cancer or hepatic metastasis are eligible to enroll, provided that, at screening, the following criteria are met:

   1. Total bilirubin is no higher than the ULN;
   2. AST and ALT are each ≤5 × the ULN;
   3. Severe liver dysfunction (Child-Pugh Class B or C) is not present; and
   4. Subjects with a history of esophageal bleeding have varices that have been sclerosed or banded and no bleeding episodes have occurred during the prior 6 months.
7. If there is a history of brain metastases treated with radiation therapy, the radiation therapy must have occurred at least 6 weeks prior to enrollment (signed ICF obtained) and the metastatic disease must have been stable since completion.
8. Willing and able to provide written Informed Consent and comply with the requirements of the study.
9. In addition, subjects enrolled in the Dose Confirmation Phase must have measurable disease, using RECIST v1.1 (Appendix 4).

Exclusion Criteria

1. Any chemotherapy, immunomodulatory drug therapy, anti-neoplastic hormonal therapy (unless it comprises androgen-deprivation therapy in a subject with prostate cancer and the dose has been stable for 3 months prior to Baseline and will remain stable during the trial), immunosuppressive therapy, corticosteroids >20 mg/day prednisone or equivalent (unless administered to prevent contrast material reactions during radiographic procedures), or growth factor treatment (e.g., erythropoietin) within 14 days prior to initiation of study drug.
2. Presence of an acute or chronic toxicity of prior chemotherapy, with the exception of alopecia or peripheral neuropathy, that has not resolved to ≤Grade 1, as determined by National Cancer Institute CTCAE v 4.0 (http://evs.nci.nih.gov/ftp1/CTCAE/About.html).
3. Positive hepatitis B virus surface antigen (HBsAg) or positive anti-hepatitis C virus (HCV) antibody.
4. Radiotherapy within 4 weeks prior to baseline.
5. Receipt of radiotherapy to >25 % of bone marrow (Appendix 5).
6. Major surgery within 28 days prior to initiation of study drug.
7. Life expectancy <12 weeks.
8. Active bacterial, fungal, or viral infection requiring systemic therapy.
9. Known human immunodeficiency virus or acquired immunodeficiency syndrome-related illness.
10. Uncontrolled congestive heart failure (New York Heart Association Classification 3 or 4, Appendix 1), angina, myocardial infarction, cerebrovascular accident, coronary/peripheral artery bypass graft surgery, transient ischemic attack, or pulmonary embolism within 3 months prior to initiation of study drug.
11. History of or ongoing cardiac dysrhythmias requiring treatment, atrial fibrillation of any grade, or persistent prolongation of the QTc (Fridericia) interval to >450 msec for males or >470 msec for females.
12. With other previous malignancies prior to study entry, except for

    1. non-basal-cell carcinoma of skin or carcinoma-in-situ of the uterine cervix
    2. the tumor was treated with curative intent more than 2 years prior to study entry.
13. Treatment with the following pharmaceutical or herbal agents within 14 days prior to study drug uptake:

    1. known to be moderate or severe inhibitors or inducers of CYP3A4 (Appendix 2).
    2. known to be sensitive or narrow therapeutic index substrates of CYP3A4, CYP2C8, CYP2C9, or CYP2C19 (Appendix 3)

    Note:
    1. For Docetaxel, Vincristine, Phenobarbital, and Aripiprazole if the washout period had been performed ≥ 30 days, the subject can be enrolled.
    2. Subject received Amiodarone will not be enrolled.
14. Use of any investigational agents within 4 weeks of baseline.
15. Pregnant or lactating female.
16. Women of childbearing potential, unless they agree to use dual contraceptive methods which, in the opinion of the principal Investigator, are effective and adequate for that subject's circumstances while on study drug and for 3 months afterward.
17. Men who partner with a woman of childbearing potential, unless they agree to use effective, dual contraceptive methods (i.e., a condom, with female partner using oral, injectable, or barrier method) while on study drug and for 3 months afterward.
18. Any severe, acute, or chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation or study drug administration, may interfere with the informed consent process and/or with compliance with the requirements of the study, or may interfere with the interpretation of study results and, in the Investigator's opinion, would make the subject inappropriate for entry into this study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-04-24 (Actual); Primary Completion 2019-01-19 (Actual); Study Completion 2019-01-19 (Actual)

PRIMARY OUTCOMES:
the dose-limiting toxicities (DLTs) and maximum tolerated dose (MTD) of daily oral MPT0E028 in subjects with advanced solid malignancies | 28 days (Cycle 1)
  Toxicity will be graded and recorded according to National Cancer Institute Common Terminology Criteria for Adverse Events - (CTCAE v4.0). The MTD of MPT0E028 is defined as the highest dose level at which less than 1/3 of subjects experience DLT during Cycle 1 and have 6 subjects in total to confirm the safety of MTD.
the pharmacokinetic (PK) profile of MPT0E028 in subjects with advanced solid malignancies | baseline; Day 1, 8, 15 of Cycle1; Day 1 and 15 of Cycle 2, 3 and 4 (each cycle is 28 days)
  PK parameters, including area under the curve, maximum plasma concentration, trough plasma concentration, time to maximum plasma concentration, apparent oral clearance, and plasma half-life will be determined.
the pharmacodynamic (PD) effects of MPT0E028 in subjects with advanced solid malignancies through the measurement of the biomarker peripheral blood mononuclear cell (PBMC) histone acetylation | baseline; Day 1, 15 of cycle1; Day 1 of Cycle 2, 3 and 4 (each cycle is 28 days)
  PBMC histone acetylation status will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Jing-Ping Liou, Study Director — Taipei Medical University
Locations (2):
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Undecided